CLINICAL TRIAL: NCT02240251
Title: A Prospective Review of Excimer Laser Assisted Inferior Vena Cava (IVC) Filter Retrieval
Brief Title: Excimer Laser Assisted IVC Filter Retrieval
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Robert Lewandowski, Primary Investigator, Northwestern University
Other Study IDs: NU STU 00058721
Record Dates: First submitted 2014-09-10; First posted 2014-09-15 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: IVC Filters
Keywords: Inferior Vena Cava Filter; IVC Filter; IVC filter removal; Excimer Laser

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing IVC filter removal using the excimer laser: Laser Assisted IVC Filter Removal
  Interventions: Other: Prospective Chart Review

INTERVENTIONS:
Other: Prospective Chart Review — The laser assisted IVC filter removal procedure itself is not part of this study. This is a prospective chart review for patients undergoing this procedure.

SUMMARY:
This is a prospective chart review to follow our laser-assisted IVC filter retrieval patients. We intend to validate existing literature and scientific findings by publishing our own clinical experience in difficult IVC filter retrievals.

DETAILED DESCRIPTION:
At Northwestern Memorial Hospital in Chicago, IL USA, IVC filters are successfully removed >95%. Technical failures, although rare, are usually related to excessive endoluminal scarring at the point of IVC filter implantation. Adjunctive (or advanced) removal techniques are often employed in difficult cases. The excimer laser sheath has been successfully used at Northwestern for patients who had failed all other retrieval techniques.

Before a patient is to undergo an IVC filter removal using the Excimer Laser Sheath they will be consented to participate in the chart review study and become a part of a registry kept at Northwestern Memorial Hospital. The procedure itself is not being used as part of the study. Chart reviews will be completed and data collected on the procedure to remove the filter. Follow up after the procedure by phone call and chart review will be completed at least once, 1 week after the filter removal.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be male and female aged 18 years to 100 years old who were treated with either permanent or retrievable IVC filter placement and were referred to the Interventional Radiology or Vascular Surgery departments for IVC filter retrieval starting December 1, 2011.
* Patients have failed all other traditional methods/attempts at removal of their IVC filter.

Exclusion Criteria:

* Patients who refuse the use of the excimer laser device to attempt to remove their IVC filter.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anyone ages 18-100 years old that will undergo laser assisted IVC filter removal at Northwestern Memorial Hospital in Chicago IL USA
Sampling Method: Non-Probability Sample
Enrollment: 535 (Actual)
Dates: Start 2012-01-03 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Evaluate any adverse events related to laser assisted IVC filter removal | up to 1 year after Laser Assited IVC filter removal
  The number and severity of adverse events will be recorded to evaluate safety. This will be conducted as a phone call to the patient 1 week after IVC filter removal and then as a chart review only.
Effectiveness of Laser Assisted IVC filter removal | At time of IVC filter removal
  Success rate of removing IVC filters using the laser will be recorded. If a filter cannot be removed with the laser the reason for this failure will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lewandowski, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States